CLINICAL TRIAL: NCT06767397
Title: Factors Influencing the Hemodynamic Stability and Its Management in Patients Undergoing Pelvic Surgery Under Spinal and General Anesthesia
Brief Title: Factors Influencing Hemodynamic Stability and Its Management in Patients Undergoing Pelvic Surgery Under Spinal and GA
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/035
Record Dates: First submitted 2024-12-18; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: general anesthesia — To evaluate the factors that affect the hemodynamic stability in patients undergoing spinal anesthesia and general anesthesia during pelvic surgery.

SUMMARY:
Patients are at risk for hemodynamic instability both during and after surgery, as it is an independent predictor of long-term patient morbidity and length of hospital stay. The development of hemodynamic instability is caused by a number of factors. When these risk factors are prevented or treated, patients may experience less hemodynamic instability during pelvic surgery, as well as the morbidity and mortality that come with it in both spinal and general anesthesia.

DETAILED DESCRIPTION:
The objective of this study was to evaluate the factors that affect the hemodynamic stability and evaluate the effectiveness of different management strategies employed to maintain hemodynamic stability during spinal and general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older.
* ASA (American Society of Anesthesiologists) physical status classification I and II.
* Patients scheduled for elective pelvic surgery.
* Can give informed consent or has a legal representative to give consent.
* There are no contraindications to spinal or general anesthesia based on preoperative assessment (e.g, severe cardiovascular disease, no previous history of adverse anesthetic reactions).

Exclusion Criteria:

* Age below 18 years.
* Emergency procedures or that require immediate intervention.
* Pregnancy or breastfeeding status.
* Conditions such as spinal cord disease and severe coagulopathy that are recognized contraindications to spinal or general anesthesia.
* ASA physical status classification III and above.
* History of severe adverse reactions to anesthesia or known allergy to anesthetic agents.
* Concurrent involvement in additional clinical trials that could have an impact on the treatment of anesthesia or hemodynamic results.
* Individuals with substantial comorbidities (such as uncontrolled hypertension or heart failure) that might complicate hemodynamic responses.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intraoperatively hemodunamic instability during spinal and general anesthesia was adressed and also evaluate its management.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic instability | 12 Months
  Hemodynamic instability determined by criteria such as fluctuations of ± 20% in the systolic or diastolic blood pressure from the baseline and measured in millimetre of mercury), fluctuations in heart rate (e.g., pulse rate ± 10% of baseline), and the lack of clinically significant hypotension or episodes of bradycardia.Oxygen saturation measured by pulse oximeter and < 90% of SPO2 was considered desaturated.
Self-designed questionnaire | 12 Months
  Self-designed questionnaire for the evaluation of the factors like Age in years, weight in kilograms, Physical health status by (ASA) American Society of Anesthesiologists classification where ASA I was physically fit patients having only surgical pathology and ASA II patient with mild systemic disease. scoring from (1-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Mardan Medical Complex, Mardan, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No